CLINICAL TRIAL: NCT02999711
Title: A Randomised, Double-blind, Placebo-controlled, Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Effects of Subcutaneously Administered REGN3500 in Adult Patients With Moderate Asthma
Brief Title: Study of Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of REGN3500 in Adults With Moderate Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R3500-AS-1619; 2016-002979-95 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Asthma; Moderate Asthma
MeSH Terms: conditions — Asthma | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): REGN3500 low dose or placebo
  Interventions: Drug: REGN3500; Drug: Placebo
- Cohort 2 (Experimental): REGN3500 medium dose or placebo
  Interventions: Drug: REGN3500; Drug: Placebo

INTERVENTIONS:
Drug: REGN3500 — REGN3500 dose
Drug: Placebo — Matching placebo

SUMMARY:
Purpose of this study is to assess the safety and tolerability of multiple ascending subcutaneous doses of REGN3500 to moderate asthmatics.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18 to 32 kg/m2
* A diagnosis of moderate asthma (according to GINA 2015) for a period of at least 2 years prior to screening.
* Patient must use a stable medium daily dose level of inhaled corticosteroids (ICS) as defined by GINA guidelines, ie, total daily dose of ICS >400 μg and ≤800 μg/day of budesonide or equivalent for at least 1 month prior to screening and during the study
* A pre-bronchodilator forced expiratory volume in the first sec (FEV1) ≥60% and ≤90% of the predicted normal values at screening and pre-dose at screening
* A documented positive response to the reversibility test at the screening, defined as improvement in FEV1 ≥12% and ≥200 mL over baseline after 400 μg salbutamol Pmdi
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent.

Key Exclusion Criteria:

* Clinically significant abnormal CBC, clinical chemistry, and urine analysis at screening.
* Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, prior to screening.
* History of life-threatening asthma
* Occurrence of asthma exacerbations or respiratory tract infections within 4 weeks prior to screening.
* Diagnosis of any other airway/pulmonary disease such as Chronic Obstructive Pulmonary Disease (COPD) as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (GOLD 2016); or other lung diseases (eg, emphysema, idiopathic pulmonary fibrosis, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency or restrictive lung disease).
* Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 1 month prior to screening.
* Use of oral antibiotics/anti-infectives within 2 weeks prior to screening.
* Known sensitivity to doxycycline or tetracyclines, or to any of the components of the investigational product formulation.
* Recent (within the previous 2 months) bacterial, protozoal, viral, or parasite infection.
* History of tuberculosis or systemic fungal diseases
* Patients treated with a monoclonal antibody based therapy (such as an anti-IgE, anti-IL-5), a biologic therapy or immunotherapy (subcutaneous immunotherapy [SCIT], sublingual immunotherapy [SLIT], or oral immunotherapy [OIT]) in the previous 12 weeks prior to screening and during the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) after repeat subcutaneous administration | Up to 36 weeks
Severity of TEAEs after repeat subcutaneous administration | Up to 36 weeks

SECONDARY OUTCOMES:
The concentration-time profile of REGN3500 after repeat subcutaneous administration | Up to 36 weeks
Immunogenicity of REGN3500 assessed by measurement of anti-drug antibodies | Up to 36 weeks
Percent change in total from baseline forced expiratory volume (FEV) at day 29 | Baseline to week 4
Percent change of the average of the prior 7 days of FEV1 at day 29 compared to average daily FEV1 during the last 14 days of screening | From -14 days screening to week 4
Absolute change from baseline fractional exhaled nitric oxide (FeNO) at day 29 | Baseline to week 4
Percent change from baseline FeNO at day 29 | Baseline to week 4
Change from baseline in biomarkers at day 29 | Baseline to week 4
Percent change from baseline in biomarkers at day 29 | Baseline to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- United Kingdom (3):
  - Regeneron Research Site, Belfast, Northern Ireland
  - Regeneron Research Site, London
  - Regeneron Research Site, Manchester

REFERENCES:
- [Derived] Kosloski MP, Kalliolias GD, Xu CR, Harel S, Lai CH, Zheng W, Davis JD, Kamal MA. Pharmacokinetics and pharmacodynamics of itepekimab in healthy adults and patients with asthma: Phase I first-in-human and first-in-patient trials. Clin Transl Sci. 2022 Feb;15(2):384-395. doi: 10.1111/cts.13157. Epub 2021 Sep 29. PMID 34523807